CLINICAL TRIAL: NCT06633185
Title: Effect of Phenytoin Cream on Wound Healing After Anal Fissure Surgery; a Randomized Controlled Trail.
Brief Title: Effect of Phenytoin Cream on Wound Healing After Anal Fissure Surgery.
Acronym: RCT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmad Sakr, principal investigator, Mansoura University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 223345
Record Dates: First submitted 2024-10-04; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-09

CONDITIONS: Anal Fissure Chronic; Anal Fissure; Wound Healing
MeSH Terms: conditions — Fissure in Ano | interventions — Phenytoin

STUDY DESIGN:
Intervention Model Description: 1st arm includes those patients who underwent application of topical phenytoin cream after anal fissure surgery, while the other arm includes those without application of any creams( control).
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Topical anal phenytoin cream application (Active Comparator): local application of phenytoin cream on anal wound post internal sphincterotomy for chronic anal fissure.
  Interventions: Drug: phenytoin cream
- control arm (Active Comparator): includes those with internal sphincterotomy but without application of topical phenytoin cream
  Interventions: Drug: no phenytoin cream

INTERVENTIONS:
Drug: phenytoin cream — application of the cream after internal anal sphincterotomy versus non application.
  Other Names: heal quick; phenytoin
  Arms: Topical anal phenytoin cream application
Drug: no phenytoin cream — Non application of the phenytoin cream
  Other Names: heal quick
  Arms: control arm

SUMMARY:
This study aims to compare the effect of phenytoin cream on wound healing after anal fissure surgery compared to control group.

DETAILED DESCRIPTION:
Introduction Anal fissure is defined as an elliptical or longitudinal tear in the anoderm distal to the dentate line, exactly proximal to or at the level of the anal verge . It is one of the most painful anal disorders that inversely affect the life quality of the patients .

Acute anal fissure is a simple rupture in the anoderm existing for less than two months and it is associated with anal pain, spasm, and/or bleeding with defecation. Chronic anal fissure is present for more than six weeks and it is characterized by exposed fibers of internal anal sphincters at the base, hypertrophied anal papilla proximally, and a skin tag or sentinel pile .

Conservative methods are likely to fail and have a higher failure rate with chronically recurring anal fissures. In these situations, the gold standard is the internal sphincterotomy. This surgical procedure treats chronic fissure by preventing hypertonia of the internal sphincter .

Wound healing is an essential step during the procedure of post-operative care after anal surgery . For example, it is believed that a desirable wound healing could help reduce the post-operative pain after hemorrhoidectomy, which quite commonly causes delayed patient discharge .

However, due to the unusual circumstance, the wound healing after anal surgery is frequently delayed by postoperative complications, such as bleeding, infection and edema, despite the use of wound healing creams . Therefore, it is still necessary to investigate more efficient therapeutic regimen to accelerate the postoperative wound healing after anal surgery.

Phenytoin is an anticonvulsant non-sedative agent, studied as a topical cream in skin lacerations, diabetic foot, pressure ulcer, and leprosy as well as oral and dental injuries . Its efficacy has been approved in all of the previous fields . This agent could activate fibroblastic proliferation, attenuate collagenase activity, inhibit glucocorticoid production, increase granulation tissue, activate angiogenesis and decrease microbial infection for accelerating wound repair .

Aim of the Work The current study will be conducted to evaluate the effect of topical phenytoin cream application on the healing process of the anal wound, following sphincterotomy for chronic anal fissure.

Patients and Methods Study design This is a prospective randomized controlled trial that will be conducted at the colorectal surgery unit of the general surgery department, at Mansoura university hospitals between January 2022 and January 2023.

Eligibility criteria Patients of both sexes, who aged between 18 and 65 years old, with chronic anal fissure after failure of previous conservative treatment including dietary modifications, laxatives, and topical therapy will be included in this study. Whereas, surgically unfit patients due to multiple comorbidities, patients with concomitant other anorectal pathology, patient with anal fissure secondary to inflammatory bowel disease, patients with active anorectal sepsis and patients with previous anal surgery will be excluded.

Random sequence generation and blinding Patients will be randomized to one of two equal groups; group I (treatment group) will be treated with lateral internal sphincterotomy with topical application of phenytoin 2% (Heal Quick®, Al hadidi pharm, Egypt), and group II (control group) will be treated with lateral internal sphincterotomy alone.

Randomization will be undertaken by the sealed envelope method using randomization software (www.randomization.com). The operating surgeon will not be aware to the nature of the study.

Preoperative assessment Detailed history will be taken from the patients with regard to complaint and its duration, associated medical conditions, previous surgical operations, previous treatments for the current condition, presence of anal pain, constipation and fecal continence state. Thorough clinical examination will be done for all patients. Local anorectal examination will be performed by direct inspection and digital rectal examination, to confirm presence of anal fissure and to exclude associated anorectal lesions. The diagnosis with chronic anal fissure was established when the patient report persistence of his symptoms for more than six weeks, along with the presence of a fissure showing the signs of chronicity (indurated edges, visible internal sphincter fibers through the base of the fissure, hypertrophic anal papilla, and sentinel pile) [14].Routine laboratory investigations including complete blood count, liver and kidney function tests, prothrombin time, and random blood glucose level will be conducted.

Operative technique:

All patients will be provided with an informed consent regarding the procedure and its complications. All patients will be placed in lithotomy position after receiving spinal anesthesia. Lateral internal sphincterotomy will be performed for all cases. The anal mucosa will be grasped using a pair of forceps, and after excision of the skin tag, the internal sphincter will be identified and separated from anal mucosa using a dissecting scissor, then a tailored internal anal sphincterotomy will be performed at 5 o'clock position by dividing the internal sphincter fibers using diathermy. After that, the wound will be left open for drainage. Proper hemostasis will be asserted then pressure dressing will be placed on the anal verge for 12 hours.

Post-operative:

Patients will be monitored in the regular ward by vital signs assessment and observation of the anal wound. Patients will be instructed to do frequent Sitz bath every six hours. During the postoperative period all patients will receive a single dose of intravenous cephalosporins and then followed by oral quinolones tablets and Non-steroidal anti-inflammatory drug (NSAIDS) for one week. For group I, additional topical phenytoin cream 2% will be commenced. It will be administered topically over wound, twice daily for one month after operation. All patients will be discharged home in the 1st postoperative day as long as there are no complications.

End points and follow up

All patients will be followed up at the outpatient clinic, every week for 1 month and the following outcomes will be assessed between both groups:

1. The primary endpoint will be the duration of healing of anal fissure. It will be defined as complete epithelization of the anal wound. Whereas, the secondary outcome will be the post-operative complications.
2. Post-operative pain according to the visual analogue scale (VAS)[15].
3. Postoperative analgesic requirements including whether the patient required additional opioids.
4. Immediate post-operative complications e.g anal bleeding or urine retention.
5. Time taken to return to daily activities in days.
6. Time taken for the patient to defecate without pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes,
* Aged between 18 and 65 years old,
* with chronic anal fissure after failure of previous conservative treatment.

Exclusion Criteria:

* surgically unfit patients due to multiple comorbidities,
* patients with concomitant other anorectal pathology,
* patient with anal fissure secondary to inflammatory bowel disease,
* patients with active anorectal sepsis
* patients with previous anal surgery .

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
The duration of healing of anal fissure. | 21 to 30 days
  The primary endpoint will be the duration of healing of anal fissure in days. It will be defined as complete epithelization of the anal wound.

SECONDARY OUTCOMES:
post operative complications and others | 14 to 21 days
  Postoperative analgesic requirements including whether the patient required additional opioids. It is measured by number of analgesic injections needed.
  Immediate post-operative complications e.g anal bleeding or urine retention. It is measured by number of cases which developed these complications Time taken to return to daily activities in days. Time taken for the patient to defecate without pain in days .

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided